CLINICAL TRIAL: NCT03739385
Title: Generations on the Move: Intergenerational Exercise and Health Promotion
Brief Title: Generations on the Move (GIB-Study): Intergenerational Exercise and Health Promotion
Acronym: GIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Oliver Faude, Professor, University of Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-01123
Record Dates: First submitted 2018-10-11; First posted 2018-11-13 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Physical Activity
Keywords: Intergenerational; Exercise; Health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study is designed as a five-armed, cluster-randomized controlled trial with a 25-week (distributed over a school year) physical exercise training intervention. After preliminary assessment (written consent, questionnaires, personal data) the institutions with their participants will be randomly assigned to either the intergenerational group (INT), the two peer-groups PGS (peer group seniors) and PGC (peer group children) or the two control groups CONS (control group seniors) or CONC (control group children). Measurements of psychological wellbeing and physical health will occur on two occasions in all five groups: before intervention start (M1) and after the intervention period (M2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Intergenerational Group (Experimental): Pre-school children and residential seniors will receive two weekly exercise training sessions lasting 45 minutes each. All exercise training sessions are conducted by professional exercise coaches and are planned in a progressive and variable manner. The training sessions focus on balance and fundamental movement skills.
  Interventions: Other: Exercise Intervention
- Peer Group Children (Active Comparator): Pre-school children will receive two weekly exercise training sessions lasting 45 minutes each. All exercise training sessions are conducted by professional exercise coaches and are planned in a progressive and variable manner. The training sessions focus on balance and fundamental movement skills.
  Interventions: Other: Exercise Intervention
- Peer Group Seniors (Active Comparator): Residential seniors will receive two weekly exercise training sessions lasting 45 minutes each. All exercise training sessions are conducted by professional exercise coaches and are planned in a progressive and variable manner. The training sessions focus on balance and fundamental movement skills.
  Interventions: Other: Exercise Intervention
- Control Group Children (No Intervention): Pre-School children will be assessed during pre-, post- and follow-up testing procedures but will receive no exercise intervention.
- Control Group Seniors (No Intervention): Residential seniors will be assessed during pre-, post- and follow-up testing procedures but will receive no exercise intervention.

INTERVENTIONS:
Other: Exercise Intervention — The training interventions of all three groups (intergenerational group, peer group seniors, peer group children) will occur under professional supervision twice a week lasting over a 25-week period with training sessions lasting 45 minutes each. Control groups (control group seniors, control group children) receive no intervention.
  Arms: Intergenerational Group; Peer Group Children; Peer Group Seniors

SUMMARY:
During the past century, major demographic changes have occurred in Europe which primarily affect the older age groups. According to the Swiss federal office of statistics, the number of senior citizens has tripled (from 5.8% to 18.0%) while the number of young adults (younger than 20 years old) has decreased from 40.7% to 20.1%. There is evidence that with increasing age, physical activity and fitness level decreases. Additionally to lower physical activity, natural aging results in a decrease of muscle strength and a modulation of afferent and efferent reflex pathways due to a slowing down of neuromuscular performance. As a consequence, there are multiple consequences on general health, disease and injury rates in the older population such as a higher risk of sustaining fall injuries. An intergenerational approach combining balance and strength promotion appears to possess great potential for fall-prevention, for satisfying physical, social and behavioral need of children and seniors as well as reducing health care costs due to increased inactivity in both age groups. No studies have examined the effects of intergenerational exercise and health programs.

DETAILED DESCRIPTION:
During the past century, major demographic changes have occurred in Europe which primarily affect the older age groups. According to the Swiss federal office of statistics, the number of senior citizens has tripled (from 5.8% to 18.0%) while the number of young adults (younger than 20 years old) has decreased from 40.7% to 20.1%. Population projections indicate a reinforcement of this population aging during the upcoming decades. There is evidence that with increasing age, physical activity and fitness level decreases. Additionally to lower physical activity, natural aging results in a decrease of muscle strength and a modulation of afferent and efferent reflex pathways due to a slowing down of neuromuscular performance. Hence, there are multiple consequences on general health, disease and injury rates in the older population such as a higher risk of sustaining fall injuries. The etiology of falls is multi-factorial comprising extrinsic / environmental factors (e.g. lighting, stairs, floor surfaces, obstructed walkways, inadequate handrails etc.) and/or intrinsic / subject-related risk factors. Two important intrinsic risk factors are deficits in static/dynamic postural control and muscular imbalance and/or weakness. Interestingly, fall rates in seniors are comparable to the ones in children caused by incomplete maturation. The risk of falling during a lifespan is a U-shaped curve, with the highest risk being during childhood and after reaching the age of 65 and older.

Many studies have been able to prove that adequate exercise training programs reduce intrinsic fall factors in seniors. Up to date, guidelines concerning fall prevention in children are limited to extrinsic factors only, and it is being postulated whether fall-preventive training programs should be included in physical education curricula. The development of effective and attractive fall-preventive intervention programs targeting intrinsic fall factors are needed in order to improve physical determinants for reducing the risk of falling in both groups. Up to date, children and seniors have been examined and trained separately to improve physical fitness parameters. An intergenerational approach combining balance and strength promotion appears to possess great potential for fall-prevention for children and seniors as well as reducing health care costs due to increased inactivity in both age groups.

Research has been able to link social-emotional competencies to early school success and the growth of academic competence during elementary school. Emotional and social skill development which are basic elements of social interactions such as the affective social competence of an individual, are developed during early childhood and should be encouraged during those stages. As children's social interactions increase in frequency and complexity, they must learn to comprehend even emotionally difficult situations, they should be able to set prosocial goals and determine effective ways to solve differences with peers as well as adults. A child's social-emotional learning should also include relationship skills. In order to build and maintain positive exchanges and satisfying relationships over time, one must acquire numerous skills such as joining others in play, initiating and maintaining conversations, cooperating, listening, and taking turns. Additionally, the attitudes as well as the forming of stereotypes against the elderly develop early and remain fairly constant, posing a strong influence on their future behavior towards others. An intergenerational setting has the potential of providing an additional challenge to a child's social-emotional learning as well as preventing prejudice against the aged. By exposing children to a new and unknown setting, they are forced to adapt socially, thus promoting their social and emotional learning abilities while positively influencing their view and attitudes towards old age. Additionally, studies examining the effects of exercise on children have confirmed that exercise has positive effects on social behavior, classroom behavior and several aspects of academic performance as well as on general health-related quality of life in children.

The aging process entails diverse and distinctive cognitive changes which are primarily influenced by environmental factors and lifestyle along with functional changes due to biological effects. The aging process increases the risk of succumbing to a variety of neurological disorders including depression, Parkinson's disease, Alzheimer's dementia and ischemic stroke. The decline in cognitive functions has been linked to a decrease in physical and social activities. As a result, quality of life starts to decline, independent living cannot be sustained, social interactions are diminished, chronic diseases such as diabetes, hypertension and higher cardiovascular risks negatively impact general health and a decline in muscular force, flexibility as well as agility and balance impacts daily activities. Decrease in cardiopulmonary function was reported to damage cerebral cortex causing central nervous system disorders, which decrease overall brain function. Both long-term research from cross-sectional studies and short-term research from randomized controlled clinical trials suggest that physical activity and fitness training influences brain structure and function positively, thus combating the aforementioned neurological disorders. Aerobic exercise has been shown to be a valid therapeutic measure to combat late-life depression and increased physical fitness is a premise for maintaining cognitive functioning as well as executive functioning in seniors.

Physical inactivity, as previously established, is one of the main causes for falls in seniors on one hand, and a protective factor for succumbing to neurological disorders in the aging process on the other hand. Programs to promote physical activity in the elderly is of great interest to combat diseases, improve quality of life and providing a social network as well as reducing risk of falling, and effective programs and methods for exercise and activity promotion in seniors are therefore of great interest and importance. To implement a successful physical activity promotion program in order to counter the effects of inactivity and achieve desirable health outcomes, the target groups must adhere to regular physical activity. Evidence suggests that physical activity promotion intervention amongst older adults are generally effective when the motivators to them are suitable such as social, individual and environmental support, and that prevention programs fail due to the lack of target group-oriented approach. To ensure that health measures reach the elderly, it is necessary to formulate messages more relevant to older people and to tailor information to their specific needs and preferences. Older seniors identify the health benefits of physical activity in terms of reducing the effects of aging and being fit to play with grandchildren and are more likely to name personal responsibility and moral obligation to maintain one's health as their motivator for participating in preventive health sports and physical activities. Motivation is a key determinant of physical activity behavior, and reports of sizeable attrition from programs of structures physical activity for older adults and from personal home-based regimens confirm that maintaining the motivation for the necessary adherence is often a challenge.

Intergenerational exercise groups possesses the potential to becoming an innovative strategy for promoting physical activity in seniors. An intergenerational approach combining balance and strength appears to possess great potential for fall-prevention, for satisfying physical, social and behavioral need of children and seniors as well as reducing health care costs due to increased inactivity in both age groups. Preliminary data indicates that intergenerational relationships affect and influence participants of exercise programs by providing motivation for seniors to exercise more regularly when children are included and to increase the seniors' self-esteem. They are an opportunity to improve social integration, tolerance, social responsibility as well as the development of social and emotional skills. Through shared physical activities in which the generations alternate their support and help, both age groups can achieve beneficial effects on psychological, social, emotional and physical factors. As aforementioned, up to date children and seniors have been examined and trained separately to improve physical fitness parameters, and no evidence exists on how intergenerational exercise programs benefit not only physical health but also social-emotional skills and psychological wellbeing. Even though no studies have examined the effects of intergenerational exercise and health programs, intergenerational approaches have been made in social, musical and artistic settings with promising preliminary outcomes in terms of mutual understanding, tolerance and social belonging. An intergenerational setting possesses the potential of providing an additional challenge to a child's social-emotional learning as well as preventing prejudice against the aged. By exposing children to a new and unknown setting, they are forced to adapt socially, thus promoting their social and emotional learning abilities while positively influencing their view and attitudes towards old age. Additionally, studies examining the effects of exercise on children have confirmed that exercise has positive effects on social behavior, classroom behavior and several aspects of academic performance as well as on general health-related quality of life in children. In regard of the aforementioned fall incidence in both age groups, a combined exercise program targeting intrinsic fall-factors (impaired static and dynamic postural control as well as deficits in muscle strength) could reduce fall-risk and in turn reduce fall-related costs.

Considering this background, the proposed study aims at comparing the effects of intergenerational exercise training compared to peer-group exercise training and control groups on parameters of psychological wellbeing and physical health. Psychological wellbeing include quality of life, fear of falling, mental health, independent living, pain, social participation and coping for seniors, while the children will be assessed on their emotional and social capabilities such as prosocial behavior, cooperation, empathy, emotional regulation and their view on aging. Physical health parameters include functional mobility, static and dynamic balance as well as cardiovascular health.

The following main research questions will be addressed:

* Do the three exercise training groups differ in adherence to exercise program?
* Do the three intervention groups differ in terms of improving psychological wellbeing?
* Do the three intervention groups differ in terms of changes in functional mobility, balance and cardiovascular health?

The research can be categorized in the risk category A according to the local ethics committee. Measurements are non-invasive and represent no risk for participants. The intervention consists of a psychological and physical health benefitting exercise programs. The study corresponds to Category A risk for activity-related adverse events are similar or lower than independent physical activity participation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy seniors of at least 65 years of age.
* Healthy children in the 2 years of kindergarten between the ages of 4 and 7 are included.

Exclusion Criteria:

* Chronic and / or congenital heart failure
* Peripheral arterial occlusive diseases

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Number of attended exercise sessions | 25 weeks intervention
  Primary outcome is adherence to the exercise intervention. Adherence corresponds to the total number of attended training sessions by each participant. Adherence will only be measured in the three intervention groups (intergenerational group, peer group seniors, peer group children).

SECONDARY OUTCOMES:
Quality of Life, AQoL-8D Score | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors is quality of life using the Assessment of Quality of Life, 8D (AQoL-8D). Scale ranges for single questions are from 1 to 5, whereby the total score is calculated by the sum of the individual scores. Lower scores represent a high quality of life, while high scores stand for low quality of life.
Independent Living | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors is Independent Living using the Assessment of Quality of Life (AQoL-8D). Scale ranges for single questions are from 1 to 5, whereby the total score is calculated by the sum of the individual scores. Lower scores represent a high independency, while high scores stand for low independency.
Mental Health | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors is Mental Health using the Assessment of Quality of Life Questionnaire (AQoL-8D). Scale ranges for single questions are from 1 to 5, whereby the total score is calculated by the sum of the individual scores. Lower scores represent good mental health while higher scores represent bad mental health.
Fear of Falling | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors is Fear of Falling using the Fall Efficacy Scale (FES). Sore ranges for individual questions range from 1 to 4, whereby the total score of all 16 questions is the total score. Low values show a low fear of falling while high scores represent a great fear of falling.
General Health | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors is General Health using the 36-Item Short Form Survey (SF 36). Answers are scored individually according to a template whereby the range is from 0 points (very low health) to 100 (excellent health). The mean value of questions represent the general health, whereby low values represent low health and high scores represent good general health.
Gait Analysis | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors is time (in seconds) needed during a 10m gait analysis.
Chair to Rise Test | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors is time (in seconds) needed to stand up and sit back down five consecutive times
Static Balance | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors is path length (mm) during a 10-second tandem balance test
Grip Force | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors and children ist force in newton (N) or in kilograms (kg) of their grip. The higher the value (N or kg), the better outcome it represents (force). Grip force will be assessed using the Automated Grip Force Assessment protocol of the Leonardo Mechanograph.
Arterial Stiffness | 1 Year (Pre- and post measurements)
  Secondary outcomes for seniors and children ist Pulse Wave Velocity (PWV)
Prosocial Behavior | 1 Year (Pre- and post measurements)
  Secondary outcomes for children ist Prosocial Behavior using the Strengths and DIfficulties Questionnaire (SDQ), filled out by their parents. Answers are rated from 1 to 2 points and the total score is the sum of the individual scores. Low total scores represent no difficulties while higher scores show difficulties.
Emotion Regulation | 1 Year (Pre- and post measurements)
  Secondary outcomes for children ist Emotion Regulation using the "Competences and Interests of Children" (KOMPIK) Questionnaire. Answers are scored on a scale of 1 to 5, whereby the mean value of individual scores represent the total score. Higher values represent a strong capacity for emotion regulation, while low scores indicate low capacity of emotion regulation.
Empathy | 1 Year (Pre- and post measurements)
  Secondary outcomes for children ist Emotion Regulation using the"Competences and Interests of Children" (KOMPIK) Questionnaire. Answers are scored on a scale of 1 to 5, whereby the mean value of individual scores represent the total score. Higher values represent a strong capacity for empathy, while low scores indicate low capacity of empathy.
Psychological Wellbeing | 1 Year (Pre- and post measurements)
  Secondary outcomes for children ist Emotion Regulation using the "Competences and Interests of Children" (KOMPIK) Questionnaire. Answers are scored on a scale of 1 to 5, whereby the mean value of individual scores represent the total score. Higher values represent high psychological wellbeing, while low scores indicate low psychological wellbeing.
Social Relationships | 1 Year (Pre- and post measurements)
  Secondary outcomes for children ist Emotion Regulation using the "Competences and Interests of Children" (KOMPIK) Questionnaire. Answers are scored on a scale of 1 to 5, whereby the mean value of individual scores represent the total score. Higher values represent a strong capacity for social relationships, while low scores indicate low capacity of social relationships.
Gross Motor Skills | 1 Year (Pre- and post measurements)
  Secondary outcomes for children are fundamental movement skills using the Test of Gross Motor Development (TGMD-2) Test Battery
Peak Power | 1 Year (Pre- and post measurements)
  Secondary outcomes for children are peak power during a single, two-legged jump on a force plate
Arterial-to-venular Ratio | 1 Year (Pre- and post measurements)
  Secondary outcomes for children is arterial-to-venular ratio assessed during static vessel analysis

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Faude, PD. Dr., Principal Investigator — Department of Sport, Exercise, and Health, University of Basel; Henner Hanssen, Prof. Dr., Study Chair — Department of Sport, Exercise, and Health, University of Basel
Locations (1):
- Department of Sport, Exercise and Health, University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No